CLINICAL TRIAL: NCT04266990
Title: Investigation of Behaviour by Dogs Prior to Human Epileptic Seizures and Potential Underlying Mechanisms. Part III: Olfactive Discriminative Ability of Dogs When Confronted With Seizure and Non-seizure Samples Part IV: Identification of Potential Biomarkers for Epilepsy in Human Sweat.
Brief Title: Olfactive Discriminative Ability of Dogs When Confronted With Seizure and Non-seizure Samples // Identification of Potential Biomarkers for Epilepsy in Human Sweat.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-10 outbreak forced us to cancel the study
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EC2019/1294
Record Dates: First submitted 2020-01-21; First posted 2020-02-12 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; Volatile Organic Components; Seizure detection; Medical detection dogs; Dog olfaction
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epilepsy patients (Experimental): Epilepsy patients admitted for clinical purposes in the EEG monitoring units at the UZ
  Interventions: Other: Planned Sweat collection; Other: Spontaneous Sweat collection
- Healthy volunteers (Active Comparator): Healthy volunteers recruited from among colleagues from the department and hospital staff
  Interventions: Other: Healthy volunteers sweat collection

INTERVENTIONS:
Other: Planned Sweat collection — Four times a day at fixed time points (9:30, 11:30, 13:30, 15:30), a researcher will ask the volunteers to wash their hands with non-scented soap and then place a sterile cotton gauze in the palm of their non-dominant hand. After 10 minutes, the gauze will be retrieved by the researcher.
  Arms: Epilepsy patients
Other: Spontaneous Sweat collection — As the patient will be under continuous monitoring, sweat and saliva samples will be also collected during and/or right after a seizure occurs if the volunteer is not holding a gauze at that time. The sweat samples will be collected by the researcher by applying a sterile gauze to the patients hands, either during or immediately following a seizure during 10 minutes.
  Arms: Epilepsy patients
Other: Healthy volunteers sweat collection — A researcher will ask the volunteers to wash their hands with non-scented soap and then place a sterile cotton gauze in the palm of their non-dominant hand. After 10 minutes, the gauze will be retrieved by the researcher. The healthy samples will be collected on the same floor of Ghent University Hospital and as close as possible to where patients reside
  Arms: Healthy volunteers

SUMMARY:
Dogs belonging to MDD will be trained and asked to discriminate between odour sweat samples from epilepsy patients associated with a seizure ("seizure sample") and samples collected when no seizure was close in time ("non-seizure sample").

The same type positive and negative sweat samples will be analysed by Florida International University using solid phase micro extraction (SPME) GC-MS to try to identify volatile organic components (VOC) specific to the samples associated with seizures.

DETAILED DESCRIPTION:
For this research, three different types of samples will be collected

1. seizure samples from patients: (S+)
2. non-seizure samples from patients : (S-)
3. samples from healthy people (H)
4. positive control samples consisting of a standard chemical mix (C+) (Only for part IV)
5. negative control samples with gauze exposed to the environment in which the samples from patients and healthy people are taken). (C-) (Only for part IV)

2.1 Collection of type a and b samples (from patients)

Sweat samples will be collected from epilepsy patients admitted for clinical purposes in the 4 EEG units at the UZ. At the time of admission, they will be asked if they agree to collaborate with the study and with their samples being taken. The patients' care is the responsibility of the staff of Ghent University Hospital. The researcher from this study will be present to collect samples in consultation with the nursing staff.

Sample collection

All the collection material will be treated with HPLC-grade methanol, and then heated to 110 degrees in an oven. The treated material will be kept in 40 ml glass vials until the collection time.

A. Planned samples:

Four times a day at fixed time points (9:30, 11:30, 13:30, 15:30), a researcher will ask the volunteers to wash their hands with non-scented soap and then place a sterile cotton gauze in the palm of their non-dominant hand. They will be asked to close the fist and keep the gauze for 10 minutes. After 10 minutes, the gauze will be retrieved by the researcher. After later analyzing the EEG readings, the samples will be marked as S+ if a seizure happened during those 10 minutes, or S- if no seizure occurred. Samples collected 24 hours before and after a seizure will not be used for further analysis.

B. Spontaneous samples

As the patient will be under continuous monitoring, sweat samples will be also collected during and/or right after a seizure occurs if the volunteer is not holding a gauze at that time. The sweat samples will be collected by the researcher by applying a sterile gauze to the patients hands, either during or immediately following a seizure during 10 minutes. The samples will be marked as S+ after confirming with the EEG reading.

2.2 Collection of type c samples (from healthy people)

In order to ensure that environmental odour is not a confounder, samples will be also collected from healthy volunteers in the same location as where samples from patients are collected. Only sweat samples will be collected from healthy volunteers.These samples are identified as healthy samples (H). Attempts to match the samples from healthy people with those from patients based age, gender and ethnicity will be made.The healthy volunteers will be recruited from among colleagues from the department and UZ staff.

The healthy samples will be collected on the same floor of Ghent University Hospital and as close as possible to where patients reside.

2.3 Sample processing.

The gauzes containing the sweat samples will be cut in 4 pieces. Two pieces will be stored in glass vials, one frozen to -20 °C and the other stored at room temperature, these samples will be sent to shipped to Florida International University. The remaining two pieces, will be shipped to Medical Detection Dogs, will be stored in sterile Falcon tubes and frozen at -20 °C.

2.4 Medical Detection Dogs sample analysis

Two dogs belonging to MDD will be asked to discriminate between seizure and non-seizure samples from patients. They will also be asked to discriminate between seizure-samples, non-seizure samples and healthy samples. The dogs will be using an 8-arms carousel. Seven samples will be placed in one arm each and one arm will remain empty.

First, dogs must be trained to recognize the hypothetical odour that is associated with epilepsy. Consequently, prior to the trial, 30 seizure samples from different patients and 120 non-seizure and healthy samples are needed for the training of the dogs

Next, 24 seizure samples from different patients and 144 non-seizure and healthy samples will be used in a double-blinded trial (24 panels with 1 seizure samples and 6 non-seizure or healthy samples). Sample size calculation is based on the assumption of a success rate of 40% to be compared with a theoretical ratio of 14.3%. A power analysis indicates that a sample size of 24 test panels is large enough to reach a power of 80% with an alpha level of 0.05 (two-sided).

2.5. Chemical analysis

Seizure samples, non-seizure samples, healthy samples and the positive and negative controls will be sent to Florida International University for SPME GC-MS analysis.

Every month for as long as the study lasts, 3 S+, 15 S-, 5 H, 1 C+ and 1 C- sample will be shipped. Analysis of the VOC profile will allow to identify potential molecules specific to the samples associated with seizures.

ELIGIBILITY:
Inclusion Criteria:

* The person will be an adult.
* The person will experience seizures implying both or either loss of conscience or incapability of interacting normally with the environment.
* Diagnostic of epilepsy confirmed by treating neurologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Answer to the question: Is possible to train Medical Detection Dogs to identify seizure-related samples using the sense of olfaction? | 8 months
  Success rate of medical detection dogs when discriminating between seizure associated and non-seizure associated samples (success rate of 40% needed to be compared with a theoretical ratio of 14.3%)
VOC Identification | 8 months
  Identification of volatile organic molecules (VOC) specific to seizure samples should they be present in human sweat

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Gent, Ghent, Belgie, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown SW, Goldstein LH. Can Seizure-Alert Dogs predict seizures? Epilepsy Res. 2011 Dec;97(3):236-42. doi: 10.1016/j.eplepsyres.2011.10.019. Epub 2011 Nov 1. PMID 22050976
- [Background] Edney AT. Dogs and human epilepsy. Vet Rec. 1993 Apr 3;132(14):337-8. doi: 10.1136/vr.132.14.337. No abstract available. PMID 8488638
- [Background] Rooney NJ, Morant S, Guest C. Investigation into the value of trained glycaemia alert dogs to clients with type I diabetes. PLoS One. 2013 Aug 7;8(8):e69921. doi: 10.1371/journal.pone.0069921. eCollection 2013. PMID 23950905
- [Background] Wells DL, Lawson SW, Siriwardena AN. Canine responses to hypoglycemia in patients with type 1 diabetes. J Altern Complement Med. 2008 Dec;14(10):1235-41. doi: 10.1089/acm.2008.0288. PMID 19040375
- [Background] Willis, C.M.., 2005. Olfactory detection of human bladder cancer by dogs: proof of principle study. Urologic Oncology: Seminars and Original Investigations, 23(3), p.217. Available at: http://linkinghub.elsevier.com/retrieve/pii/S1078143905000323.
- [Background] Schmidt K, Podmore I. Current Challenges in Volatile Organic Compounds Analysis as Potential Biomarkers of Cancer. J Biomark. 2015;2015:981458. doi: 10.1155/2015/981458. Epub 2015 Mar 30. PMID 26317039